CLINICAL TRIAL: NCT07052019
Title: Pain Perception and Anxiety With Virtual Reality Distraction Versus Tell-Show-Do Technique in Restorative Treatment for Children With Molar Incisor Hypomineralization: A Pilot Crossover Randomized Clinical Trial
Brief Title: Pain Perception and Anxiety With Virtual Reality vs Tell-Show-Do in Children With MIH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Saleem Mojahed Abou-Musallam, Lecturer Assistant at Pediatric Dentistry Department, Cairo University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U Cairo Hagar
Record Dates: First submitted 2025-06-18; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: Molar Incisor hypomineralization; MIH; virtual reality; behavioral; pain; anxiety
MeSH Terms: conditions — Molar Hypomineralization; Behavior; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Virtual Reality then Tell-Show-Do (Experimental): Children receive restorative treatment with Virtual Reality distraction during the first session, and Tell-Show-Do technique during the second session (after washout period).
  Interventions: Device: Virtual Reality Distraction; Behavioral: Tell-Show-Do Technique
- Arm B: Tell-Show-Do then Virtual Reality (Active Comparator): Children receive restorative treatment with Tell-Show-Do technique in the first session, and Virtual Reality distraction in the second session (after washout period).
  Interventions: Device: Virtual Reality Distraction; Behavioral: Tell-Show-Do Technique

INTERVENTIONS:
Device: Virtual Reality Distraction — Children wear virtual reality glasses during restorative dental treatment to reduce pain and anxiety.
Behavioral: Tell-Show-Do Technique — Conventional behavioral technique where the dentist tells, shows, and then performs the procedure to reduce anxiety and build cooperation.

SUMMARY:
This pilot crossover randomized clinical trial aims to compare the effect of distraction using Virtual Reality (VR) versus the Tell-Show-Do (TSD) technique on pain perception and anxiety in children aged 6-12 with Molar Incisor Hypomineralization (MIH) undergoing restorative dental treatment.

DETAILED DESCRIPTION:
Molar Incisor Hypomineralization is a prevalent developmental condition affecting the enamel of first permanent molars and, occasionally, incisors. It presents significant clinical challenges due to the hypersensitivity and increased pain perception in affected teeth, which can make restorative treatment especially distressing for pediatric patients. Children with MIH are often apprehensive toward dental procedures, resulting in higher levels of dental anxiety that can impact their cooperation and the overall success of treatment. The management of pain and anxiety during restorative treatments is therefore crucial, particularly in this vulnerable population.

Behavioral management techniques, such as the Tell-Show-Do (TSD) approach, have been widely used in pediatric dentistry to alleviate anxiety and improve patient cooperation. However, recent advances in digital technology, particularly Virtual Reality (VR), offer novel, immersive forms of distraction that could enhance pain management by shifting the child's attention away from the dental procedure. VR distraction has shown promise in reducing anxiety and pain perception across various medical and dental settings, but its efficacy compared to traditional behavioral techniques, such as TSD, remains under-explored, especially in the context of MIH.

A recent systematic reviews of behavioral interventions in pediatric dentistry highlighted a lack of robust evidence regarding the effectiveness of VR as a distraction technique in dental settings, particularly in randomized controlled trials (RCTs). The reviews specifically called for more rigorous studies to directly compare VR with established techniques like TSD in managing dental anxiety and pain perception. Given this identified gap in the literature, this study aims to address these limitations by conducting a crossover randomized clinical trial to compare VR distraction with TSD in children with MIH undergoing restorative treatment. By examining both pain perception and anxiety levels, this study seeks to contribute valuable insights into the comparative effectiveness of VR and TSD, providing evidence-based recommendations for pediatric dental practitioners.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 6-12 years.
* Patients with two First Permanent molars diagnosed with MIH indicated for class I cavities.
* A cooperative and compliant patient/ parent.
* Patients not allergic to medicaments necessary to complete the procedure.
* Patients with no history of chronic systemic diseases.

Exclusion Criteria:

* MIH-affected molars require apexogenesis, apexification, regeneration or RCT.
* Non-restorable tooth.
* Previous restorative treatment.
* Periodontally affected.
* Children having systemic disease, an emotional behavioural or learning disorder.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain perception | Immediately before treatment (baseline), during treatment (within session), and immediately after treatment (post-procedure)
  Tool: Wong Baker Faces Pain Rating Scale Unit: Score 0-10

SECONDARY OUTCOMES:
Anxiety level | Immediately before treatment (baseline), during treatment (within session), and immediately after treatment (post-procedure)
  Tool: Modified Child Dental Anxiety Scale (MCDAS-f) Unit: Score 8-40
Heart Rate | Baseline (5 minutes before session), during treatment (real-time), and immediately post-treatment (within 5 minutes)
  Tool: Pulse Oximeter Unit: Beats per minute
Oxygen Saturation | Baseline (5 minutes before session), during treatment (real-time), and immediately post-treatment (within 5 minutes)
  Tool: Pulse Oximeter Unit: %

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Cairo university, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes